CLINICAL TRIAL: NCT06607783
Title: A Multi-Centre, Pivotal Stage, Study to Determine the Between MRI Scanner Reproducibility of Gold Standard Phantom Calibrated Acquisition Replicator (CARE) for Measurement of Apparent Diffusion Coefficients in the Prostate of Patients With MR Positive Lesions Destined for Biopsy
Brief Title: PRostate Cancer Enhanced Diagnosis by Calibration Technology
Acronym: PREDICT
Status: Not yet recruiting | Type: Observational
Sponsor: Gold Standard Phantoms (Industry)
Collaborators: Bioxydyn Ltd, Manchester (Unknown); National Cancer Imaging Translational Accelerator (Unknown); University College London Hospitals (Other); National Hospital of Neurology and Neurosurgery, Queens Square, London, UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: GSP001; 10071751 (Other Grant/Funding Number: Innovate UK); 340447 (Other: IRAS Project ID)
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancers
Keywords: MRI; Calibration; Prostate Cancer; Quantitative Imaging Biomarker; Reproducibility; Data interoperability; Phantom; Apparent Diffusion Coefficient; ADC; PIRAD; Diagnosis; Biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Group Males: Men with clinically suspected prostate cancer and referred for prostate MRI with Likert/PIRADS 3 or above and prior decision made to perform targeted biopsy.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Standard MRI using phantom.

SUMMARY:
The CARE® Phantom system is a medical device system that is being developed has been designed to enable the quantitative measurement of the apparent diffusion coefficient (ADC) in the prostate of patients undergoing a multi-parametric MRI (mpMRI) scan to detect prostate cancer. The final device system will comprise three elements: a calibration mat containing phantoms and embedded monitoring software, a docking station to transfer data from the phantoms, and software as a medical device (SaMD) for calibrating the resulting mpMRI images.

In this clinical trial, patients will undergo MRI scanning in different scanners using the GSP Phantoms to provide mpMRI images and phantom data for subsequent in silico analysis. The captured images and data will be used to further develop and calibrate the GSP prototype SaMD part of the medical device system, and to establish the degree of optimised reproducibility that can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years and older undergoing investigations for PCa.
* Standard of Care MRI conducted.
* One or more lesions with a Likert score of 3 or above identified on clinical reports.
* Planned targeted biopsy within 6 months from the date of clinical care MRI.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Prostate specific antigen (PSA) level > 20ng/ml within 6 months
* Previous diagnosis of prostate cancer
* Ongoing hormone treatment within 3 months prior to MRI, excluding antiandrogens or 5-alpha reductase inhibitors
* Contraindication to MRI scan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male participants with suspected prostate cancer residing in the London area.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the Reproducibility of GSP CARE Reference Phantom on Different MRI Scanners | From date of first participant enrolment until the date of the final ADC measurement analysis, assessed up to 18 months.
  To determine the reproducibility of GSP CARE reference phantom corrected lesion ADC measurements when the phantom is used on different MRI scanners for measurement of ADC in prostate.
  Voxel-wise median ADC values will be obtained for each lesion region of interest (ROI), referred to in the synopsis as "ADC measurements".
  The study is designed for 3 pairwise comparisons of 3 MRI scanners, enabling reproducibility determination between each pair of scanners. The study is powered for each pairwise comparison, based on a single lesion per patient.

SECONDARY OUTCOMES:
Assessment of Reproducibility Between MRI Scanners | From date of first participant enrolment until the date of the final ADC measurement analysis, assessed up to 18 months.
  To determine whether increasing the between scanner reproducibility enables sufficiently precise voxelwise median ADC measurements (i.e. variance is not inferior to a minimally acceptable variance) to be able to distinguish between the expected ADC values from clinically significant and clinically insignificant prostate lesions.
Observation of the Extent to Which Biopsy Can be Avoided when Using GSP CARE Phantom System | From date of first participant enrolment until the date biopsy results of participants are received, assessed up to 6 months.
  To investigate the proportion of men who would receive a correct clinical recommendation that biopsy could be avoided using ADC measurements with and without GSP CARE reference phantom correction. This is a feasibility analysis to indicate data needed to power a trial to demonstrate a difference in proportion. Data will be presented graphically, with 95% confidence intervals using Wilson method. The study is not powered to show a statistical significance. Comparison of paired proportions within patient of recommendations using ADC measurements with and without GSP CARE reference phantom correction.
Determination of Per-Lesion Diagnostic Accuracy of GSP CARE-Corrected ADC Measurements | From date of first participant enrolment until the date of the final ADC measurement analysis, assessed up to 18 months.
  To determine per-lesion diagnostic accuracy of ADC measurements, corrected using the GSP CARE reference phantom, for significant cancer in men scheduled for standard of care biopsy with Likert/PIRADS 3 or above scored MRI lesions. Sensitivity and specificity will be calculated per lesion, with 95% confidence intervals using Wilson method. Statistical significance will be based on 95% confidence intervals.
Determination of the Association Between GSP CARE Reference Phantom Corrected Lesion ADC Measurements and Tumour Gleason Grade | From date of first participant enrolment until the date of the final ADC measurement analysis, assessed up to 18 months.
Investigation of Device Usability | From date of first participant enrolment until the date all radiographers and participants have completed a Usability Questionnaire, assessed up to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data generated is going to be used for optimising development of Software as a Medical Device and for assessment of reproducibility.